CLINICAL TRIAL: NCT02591316
Title: Lifestyle Factors, Inflammation, and Cognition in Breast Cancer Survivors
Brief Title: Nutrition, Physical Activity, and Cognition in Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Texas State University, San Marcos (Other)
Responsible Party: Principal Investigator, Krystle Zuniga, Assistant Professor, Texas State University, San Marcos
Other Study IDs: 2014T34
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Cognitive Impairment; Cognition
Keywords: nutrition; physical activity; breast cancer survivor; cognition
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast cancer survivor: Inclusion criteria: Female breast cancer survivors (30-70yrs of age) that have completed primary treatment (chemotherapy, radiation therapy or both) within past 60 months
  Interventions: Other: no intervention
- Control: Females (30-70yrs of age) with no previous cancer diagnosis.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The purpose of this study is to examine the relationship between nutrition, physical activity and brain function in breast cancer survivors.

DETAILED DESCRIPTION:
The current study will examine the potential relationships between physical activity, dietary intake, body composition and cognition in breast cancer cancer survivors and age-matched women without a previous cancer diagnosis. Additionally, we will measure blood inflammatory markers to explore the relationship between lifestyle factors and inflammation.

The study involves two, 1hr appointments at Texas State University. The first visit will include cognitive testing and body composition assessment. Participants will be given an activity monitor to wear for one week and a packet of questionnaires to complete at home. At the second visit, a fasted blood sample will be collected, and participants will complete a food frequency questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivors must have completed primary treatment (chemotherapy, radiation therapy or both) within past 60 months
* age-matched controls must have no previous cancer diagnosis
* Female
* no history of stroke, heart attack or transient ischemic attack
* not currently pregnant; can speak, read, and write English
* can attend all testing sessions
* not blind or legally blind; nonsmoker
* no current use of computer-based brain training games (e.g. Lumosity ®, BrainHQ ®).

Exclusion Criteria:

* male
* < 30 or > 70 years of age
* breast cancer survivor > 60 months from last treatment or currently undergoing primary treatment
* breast cancer survivor never treated with chemotherapy and/or radiation
* previous cancer diagnosis other than breast cancer

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female breast cancer survivors and women who have never had a previous cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cognition | Baseline
  A series of computer-based cognitive tasks will be administered via the NIH Toolbox Cognition Battery

SECONDARY OUTCOMES:
Physical Activity | Baseline
  Physical activity will be measured by a waist-worn accelerometer
Diet Quality | Baseline
  Diet will be assessed by completion of the online-administered 2005 Block Food Frequency Questionnaire
Body Composition (objectively measured) | Baseline
  Body composition will be evaluated by BOD POD assessment
Inflammatory Markers | Baseline
  A fasted blood sample will be collected for measurement of inflammatory markers

OTHER OUTCOMES:
Medical History | Baseline
  Self-reported medical history
Quality of Life | Baseline
  Series of questionnaires assessing various aspects of quality of life including physical and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Krystle E Zuniga, PhD, RD, Principal Investigator — Texas State University, San Marcos
Locations (1):
- Texas State University, San Marcos, Texas, United States